CLINICAL TRIAL: NCT06181123
Title: Comparison of Functionality, Physical Activity, Cardiac and Respiratory Parameters Between Patients With Mood Disorders and Healthy Controls
Brief Title: Cardiopulmonary Assesments in Mood Disorders
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Irem Hüzmeli, assistant professor, Mustafa Kemal University
Other Study IDs: Mustafa Kemal University
Record Dates: First submitted 2023-11-29; First posted 2023-12-26 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Mood Disorders; Physical Inactivity; Respiratory Function Impaired
MeSH Terms: conditions — Mood Disorders; Sedentary Behavior; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy group: Demographic data, clinical characteristics, exercise capacity (6 MWT, 3 min. Step test), functionality (vertical jump test, functional reach test), respiratory parameters (Respiratory muscle strength, pulmonary function test, MMRC scale), physical activity level (IPAQ, short form).
  Interventions: Other: Cardiorespiratory Assesments
- Patient group: Demographic data, clinical characteristics, exercise capacity (6 MWT, 3 min. Step test), functionality (vertical jump test, functional reach test), respiratory parameters (Respiratory muscle strength, pulmonary function test, MMRC scale), physical activity level (IPAQ, short form).
  Interventions: Other: Cardiorespiratory Assesments

INTERVENTIONS:
Other: Cardiorespiratory Assesments — The following were evaluated to make comparisons between the two groups: Demographic data, clinical characteristics, exercise capacity (6 MWT, 3 min. Step test), functionality (vertical jump test, functional reach test), respiratory parameters (Respiratory muscle strength, pulmonary function test, MMRC scale), physical activity level (IPAQ, short form).
  Other Names: assesments

SUMMARY:
The importance of cardiorespiratory impact in mental diseases is generally emphasized in studies, but it is noteworthy that cardiorespiratory affects in mood disorders have not been sufficiently investigated. This study aims to compare individuals with mood disorders and healthy people in terms of exercise capacity, functionality, respiratory muscle strength, respiratory functions, dyspnea and physical activity level.

DETAILED DESCRIPTION:
The cross-sectional study was carried out with 30 patients with diagnosis of mood disorder who applied to the Hatay Mustafa Kemal University Research and Practice Hospital, Mental Health and Diseases clinic, and 35 healthy individuals whose age, gender were matched. Clinical characteristics, exercise capacity (6-minute walking test, 6MWT; 3-minute Step test, 3MST), functionality (vertical jump test, functional reach test), respiratory parameters (Respiratory muscle strength, pulmonary function test), dyspnea (Modified Medical Research Council, MMRC scale), physical activity level (short form international physical activity questionnaire, IPAQ) was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who had undergone a general physical examination in the past 6 month
* reported being free of significant cardiovascular, respiratory, neuromuscular, and endocrine disorders that preclude safe participation

Exclusion Criteria:

* Individuals with significant cardiovascular, neuromuscular and endocrine disorders,
* pregnant women,
* people under 18 years old
* disabled individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * being over 18 years of age
  * being diagnosed with mood disorders
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Six minute walking test (Evaluation of exercise capacity) | Baseline
  Six minute walking test, The patients were allowed to rest for at least 30 minutes pre-starting the test, which was performed according to ATS criteria. The participants were asked to walk as fast as they can without running in a 30-meter straight corridor for 6 minutes at their own walking pace
3 minute step test (Assessment of exercise capacity) | Baseline
  3 minute step test, In this test, the person ascends and descends the 30.5 cm step with the rhythm of the metronome set at 96 beats/min for 3 minutes.

SECONDARY OUTCOMES:
Vertical jump test (Functionality 1) | in a time through the study completion, an average of 5 minutes
  Vertical jump test, The vertical jump test is used to evaluate performance characteristics. The person to be tested lies on a flat platform as far as he can with one arm, placing equal weight on both extremities, and is marked. Then, the person jumps and the last point he can reach by jumping is marked. Applying these procedures, the difference between the two marked points was recorded .
Forced vital capacity (FVC) (Pulmonary function) | Baseline
  Pulmonary function test was performed with a portable spirometer (SPIROBANK II® USA). Forced vital capacity (FVC). The test was performed in the sitting position. The best of the 3 maneuvers that were technically acceptable and had 95% agreement with each other was selected for statistical analysis.
forced expiratory volume in the first second (FEV1) (Pulmonary function) | Baseline
  Pulmonary function test was performed with a portable spirometer (SPIROBANK II® USA). forced expiratory volume in the first second (FEV1)
ratio of forced expiratory volume in the first second to forced vital capacity (FEV1/FVC) | Baseline
  Pulmonary function test
peak expiratory flow rate (PEF) | Baseline
  Pulmonary function test
forced mid-expiratory flow rate (FEF25-75%) | Baseline
  Pulmonary function test
Respiratory muscle strenght | Baseline
  Respiratory muscle strength was evaluated using a portable, electronic oral pressure measurement device (MicroRPM, Micro Medical England) according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. Respiratory muscle strength was evaluated with an oral pressure device that gives MIP MEP results. If the difference was greater than 5% or 5 cmH2O between the two best measured values, the measurement was repeated, and the best values for the analyses were kept.
Physical activity | Baseline
  The physical activity level was evaluated using the short form of the International Physical Activity Questionnaire (IPAQ) (21). IPAQ consists of seven questions in total.
The Functional Reaching Test (Functionality 2) | Baseline
  In the Functional Reaching Test, another functionality test, the individual approaches the wall in a sideways position with shoulder facing the wall. Then, the individual opens the feet at shoulder level and clasps the hand, bringing it to a 90-degree flexion position. The part where the 3rd metacarpal bone of the hand meets the wall is marked. The participant is asked to lie forward as much as possible without breaking the contact of the heels with the ground and without taking a step. Then, the distance between this starting and ending point is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Görgün, student, Study Director — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Merkez, Turkey (Türkiye)